CLINICAL TRIAL: NCT05480007
Title: Effect of DPP-4I and Related Treatment on Non-alcoholic Fatty Liver Disease
Brief Title: Non-alcoholic Fatty Liver Disease and Its Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 085348
Record Dates: First submitted 2022-07-24; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): did not take medicine
- DPPVI (Experimental): received sitagliptin treatment (100mg per day)
  Interventions: Drug: Sitagliptin
- metformin (Experimental): received metformin (500mg three times per day)
  Interventions: Drug: Metformin
- metformin +DPPVI (Experimental): received sitagliptin (100mg per day) and metformin (500 mg three times per day)
  Interventions: Drug: sitagliptin and metformin

INTERVENTIONS:
Drug: sitagliptin and metformin — sitagliptin plus metformin group who received sitagliptin (100mg per day) and metformin (500 mg three times per day) (20 patients)
  Other Names: DPP
  Arms: metformin +DPPVI
Drug: Sitagliptin — sitagliptin treatment (100mg per day)
  Arms: DPPVI
Drug: Metformin — metformin group who received metformin (500mg three times per day)
  Arms: metformin

SUMMARY:
Dipeptidyl peptidase-4 inhibitors (DPP-4I), key regulators of the actions of incretin hormones, exert anti-hyperglycemic effects in type 2 diabetes mellitus (T2DM) patients. A major unanswered question concerns the potential ability of DPP-4I to improve intrahepatic lipid (IHL) content in nonalcoholic fatty liver disease (NAFLD) patients. The aim of this study was to evaluate the effects of sitagliptin on IHL in NAFLD patients.

DETAILED DESCRIPTION:
A prospective, 24-week, single-center, open-label, comparative study enrolled 68 Chinese NAFLD patients with T2DM. Subjects were randomly divided into 4 groups: control group who did not take medicine (14 patients); sitagliptin group who received sitagliptin treatment (100mg per day) (17 patients); metformin group who received metformin (500mg three times per day) (17 patients); and sitagliptin plus metformin group who received sitagliptin (100mg per day) and metformin (500 mg three times per day) (20 patients). IHL, physical examination (waist circumstances, WC; body mass index, BMI), glucose-lipid metabolism (fasting plasma glucose, FPG; hemoglobin A1c, Hb1A1c; triglycerides; cholesterol; alanine aminotransferase, ALT; aspartate aminotransferase, AST) were measured at baseline and at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 30-70 years old
* fulfillment of the diagnostic criteria for T2DM by WHO in 1999 (HbA1c ranged from 7% to 10%, FPG < 11 mol/l, 2-hour blood glucose postprandial < 20mmol/l)
* Fulfillment of the diagnostic criteria for NAFLD according to the guidelines of the Chinese Medical Association in 2010. The IHL content was measured by using 1H-magnetic resonance spectroscopy (1H-MRS) quantitative detection, and the liver fat content of the enrolled subjects was more than 5.5%. The subjects included in this study had either no history of alcohol consumption or their alcohol intake was less than 70 g/week in males and less than 140 g/week in females. Liver transaminase and serum creatinine were less than two times the upper limit of normal

Exclusion Criteria:

* T2DM complicated with ketoacidosis, hyperosmolarity, acute and chronic infection ● serious heart, liver, kidney, lung disease, and liver damage
* alcoholic fatty liver
* drug use that influences glucose metabolism such as thiazide diuretics and hormones within three months
* Hypertension ≥ 180/110 mmHg
* gastrointestinal disease or absorption dysfunction
* recent trauma, surgery, or other conditions resulting in an increased stress response within the past three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01-30 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
intrahepatic lipid (IHL) | 24weeks
  hepatic steatosis

REFERENCES:
- [Derived] Wang X, Zhao B, Sun H, You H, Qu S. Effects of sitagliptin on intrahepatic lipid content in patients with non-alcoholic fatty liver disease. Front Endocrinol (Lausanne). 2022 Aug 22;13:866189. doi: 10.3389/fendo.2022.866189. eCollection 2022. PMID 36072931